CLINICAL TRIAL: NCT07045181
Title: Interpretable Prediction of Pancreatic Neoplasms in Chronic Pancreatitis Patients With Focal Pancreatic Lesions Based on XGBoost Machine Learning and SHAP
Brief Title: Prediction Model of Pancreatic Neoplasms in CP Patients With Focal Pancreatic Lesions
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: IPNPM
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pancreatitis; Pancreatic Neoplasm; Machine Learning
Keywords: Pancreatic neoplasm; chronic pancreatitis; machine learning; SHAP
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pancreatic neoplasm group: This cohort consists of chronic pancreatitis patients whose focal pancreatic lesions were diagnosed as pancreatic neoplasm
  Interventions: Diagnostic Test: XGBoost machine learning
- Non-pancreatic neoplasm group: This cohort consists of chronic pancreatitis patients whose focal pancreatic lesions were diagnosed as benign lesions
  Interventions: Diagnostic Test: XGBoost machine learning

INTERVENTIONS:
Diagnostic Test: XGBoost machine learning — XGBoost is a powerful machine learning algorithm known for its efficiency and performance. It is an optimized gradient boosting library designed to be highly efficient, flexible, and portable. XGBoost works by combining multiple weak prediction models, typically decision trees, to produce a strong predictive model. It supports various objective functions and evaluation metrics, making it suitable for a wide range of tasks, including classification and regression. XGBoost also includes features like regularization to prevent overfitting and can handle missing data effectively.

SUMMARY:
This study aims to develop XGBoost machine learning model to predict pancreatic neoplasms in CP patients with focal pancreatic lesions.

DETAILED DESCRIPTION:
Pancreatic neoplasms include various types, with pancreatic cancer being the most common and having a poor prognosis. Chronic pancreatitis (CP) can progress to pancreatic cancer, and detecting neoplasms in CP patients is challenging due to similar imaging and clinical presentations. Current diagnostic methods like CT and tumor markers have limitations, and endoscopic ultrasound-guided tissue acquisition has moderate sensitivity. Machine learning (ML) shows promise in medical fields, but its "black box" nature limits its application. SHapley additive exPlanations (SHAP) can provide intuitive explanations for ML models. This study aims to develop an ML model to predict pancreatic neoplasms in CP patients with focal pancreatic lesions and use SHAP to explain the model, aiding future research.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pancreatitis
* Patients has indeterminate focal pancreatic lesions discovered through contrast-enhanced CT scans

Exclusion Criteria:

* Patients had incomplete clinical data
* Patients had no surgical pathology results for the focal pancreatic lesions and loss to follow-up, indicating that a final diagnosis of the focal pancreatic lesions could not been established

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic pancreatitis patients who has indeterminate focal pancreatic lesions discovered through contrast-enhanced CT scans
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | 10 years
  The diagnostic yield of XGBoost machine learning, including AUC、Sensitivity、Specificity

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkegard J, Mortensen FV, Cronin-Fenton D. Chronic Pancreatitis and Pancreatic Cancer Risk: A Systematic Review and Meta-analysis. Am J Gastroenterol. 2017 Sep;112(9):1366-1372. doi: 10.1038/ajg.2017.218. Epub 2017 Aug 1. PMID 28762376
- [Background] Hao L, Zeng XP, Xin L, Wang D, Pan J, Bi YW, Ji JT, Du TT, Lin JH, Zhang D, Ye B, Zou WB, Chen H, Xie T, Li BR, Zheng ZH, Wang T, Guo HL, Liao Z, Li ZS, Hu LH. Incidence of and risk factors for pancreatic cancer in chronic pancreatitis: A cohort of 1656 patients. Dig Liver Dis. 2017 Nov;49(11):1249-1256. doi: 10.1016/j.dld.2017.07.001. Epub 2017 Jul 15. PMID 28756974
- [Background] Korpela T, Udd M, Mustonen H, Ristimaki A, Haglund C, Seppanen H, Kylanpaa L. Association between chronic pancreatitis and pancreatic cancer: A 10-year retrospective study of endoscopically treated and surgical patients. Int J Cancer. 2020 Sep 1;147(5):1450-1460. doi: 10.1002/ijc.32971. Epub 2020 Apr 3. PMID 32162688